CLINICAL TRIAL: NCT06018493
Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Essential Hypertension: a Drug Naive Randomized Controlled Trial (PARADISE-HTN-II)
Brief Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Essential Hypertension (PARADISE-HTN-II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Jiangning Hospital of Nanjing Medical University (Other); Suzhou Municipal Hospital (Other); The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Xiangqing Kong, Head of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARADISE-HTN-II
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases
Keywords: Hypertension; Cardiovascular disease; Focused ultrasound; Novel method
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, and sham-control study. The ratio of the intervention group versus sham-control group is 1:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: The masking range includes participants, most researchers (including the study leader; subjects screening researchers; follow-up researchers; sonographers; MR scanners, members of the clinical endpoint identification committee,and etc.) except for the study statistical analysts and the therapy operators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In intervention group, participants will receive the whole peri-renal fat modification therapy (including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting and initiating) Intervention: Device: focused power ultrasound mediate inferior perirenal adipose tissue modification
  Interventions: Device: focused power ultrasound mediate inferior perirenal adipose tissue modification
- sham-control group (Sham Comparator): In sham control group, participants will receive the sham control therapy(including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting),however,without initiating the focused ultrasound equipment.
  Intervention: Device: sham-control group
  Interventions: Device: sham-control group

INTERVENTIONS:
Device: focused power ultrasound mediate inferior perirenal adipose tissue modification — This novel focused power ultrasound is an externally delivered, completely noninvasive focused therapeutic ultrasound device. It is capable of focusing the resulting ultrasound beam to a small "cigar"-shaped volume and monitoring the temperature of the target area, which leads to the rapid elevation of the peri-renal adipose tissue temperature and the destruction of target tissue eventually.
  Arms: intervention group
Device: sham-control group — participants will receive the sham control therapy(including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting),however,without initiating the focused ultrasound equipment.
  Arms: sham-control group

SUMMARY:
This randomized, blinded, sham-control trial aims to evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for essential hypertension.

DETAILED DESCRIPTION:
The increase of visceral fat is closely related to the occurrence of hypertension, and it is one of the main independent risk factors of hypertension. Visceral fat has been recognized as an important endocrine organ, and a variety of factors secreted by visceral fat lead to an increased risk of cardiovascular disease. Peri-renal fat is a special type of visceral fat which is different from other type of visceral fat in histology, physiology, and functions. The positon of peri-renal fat is more stable than other visceral fat, which might be influenced by breath or body position changes.Studies have found that perirenal fat is an early predictor of ASCVD, and its accumulation is closely related to the occurrence and development of ASCVD. Therefore, the reduction or modification of visceral fat,especially peri-renal fat , has a sufficient scientific basis for the treatment of hypertension.

In our previous experiments, this novel focused power ultrasound can rapidly and efficiently promote the perirenal adipose tissue fibrosis and control the blood pressure in the model of swine. Moreover, the investigators performed a single arm, small sample study to investigate the feasibility of the novel focused power ultrasound to modify the inferior perirenal adipose tissue in human volunteers, showing that this kind of method was feasible and safe.

In this study, the investigators aim to further evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with office systolic blood pressure (SBP) ≥ 140 mmHg and <160 mmHg, and diastolic blood pressure<100mmHg when not taking antihypertensive drugs for at least 1 month;
2. Individual with 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP≥130 mmHg；
3. The anteroposterior, transverse and axial diameters of inferior perirenal fat pad measured by ultrasound should be at least 20mm；
4. Individual is willing to sign the informed consent of the study.

Exclusion Criteria:

1. Individual with office systolic blood pressure (SBP) ≥ 160 mmHg and/or office diastolic blood pressure(DBP)≥ 100mmHg;
2. Individual diagnosed as secondary hypertension (e.g. renal parenchymal hypertension, renal artery stenosis, primary aldosteronism, pheochromocytoma, Cushing's syndrome, aortic coarctation, obstructive sleep apnea hypopnea syndrome)；
3. Individuals with ≥ 3 cardiovascular risk factors (male>55 years old, female>65 years old; smoking or passive smoking; 2-hour postprandial blood glucose 7.8-11mmol/L and/or impaired fasting glucose (6.1-6.9mmol/L); LDL-C ≥ 3.4mmol/L (130mg/dl), HDL-C<1.0mmol/L (40mg/dl) or TC ≥ 5.2mmol/L (200mg/dl); Family history of early onset of cardiovascular disease, age of onset of first degree relatives<50 years old; Abdominal obesity, waist circumference: male≥90cm, female≥85cm or BMI≥28kg/m2) or hypertensive target organ damage;
4. Individuals taking other medications that may affect blood pressure (such as glucocorticoids);
5. Individual with history of kidney or kidney surrounding tissue surgery;
6. Individuals with impairment of liver or kidney function (ALT, AST or creatinine greater than 2 times of the upper limit of normal reference);
7. Individual with myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack within 6 months of enrollment;
8. Individual with type 1 diabetes or uncontrolled type 2 diabetes；
9. Individual with uncontrolled thyroid dysfunction;
10. Individual with urinary calculi or hematuria；
11. Individual with atrial fibrillation;
12. Individual with severe structural heart disease (e.g. valvular heart disease, cardiomyopathy, congenital heart disease);
13. Individual with second degree and above atrioventricular block and/or sick sinus syndrome;
14. Individual with abnormal coagulation function;
15. Individual with infected waist skin;
16. Individual with malignant tumor;
17. Individual is pregnant, nursing or planning to be pregnant;
18. Individual is unwilling to sign informed consent;
19. Individual fails to complete the screening period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | From baseline to 1 month post-procedure
  Changes of mean systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 1-month compared with baseline

SECONDARY OUTCOMES:
Ambulatory Blood Pressure | From baseline to 3 month post-procedure
  Changes of mean systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 3-month compared with baseline
Office Systolic Blood Pressure | From baseline to 1 month post-procedure
  Changes of office systolic blood pressure at 1-month compared with baseline
Office Systolic Blood Pressure | From baseline to 3 month post-procedure
  Changes of office systolic blood pressure at 3-month compared with baseline
Ambulatory Blood Pressure | From baseline to 1 month post-procedure
  Changes of mean diastolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 1-month compared with baseline
Ambulatory Blood Pressure | From baseline to 3 month post-procedure
  Changes of mean diastolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 3-month compared with baseline

OTHER OUTCOMES:
Safety evaluation | From baseline to 3 month post-procedure
  Any severe adverse events (SAE) related to intervention. The SAE were defined as acute renal failure, acute intestinal perforation, and thromboembolic events, et al.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital/The Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Jiangning Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayashi T, Boyko EJ, Leonetti DL, McNeely MJ, Newell-Morris L, Kahn SE, Fujimoto WY. Visceral adiposity is an independent predictor of incident hypertension in Japanese Americans. Ann Intern Med. 2004 Jun 15;140(12):992-1000. doi: 10.7326/0003-4819-140-12-200406150-00008. PMID 15197016
- [Background] Chandra A, Neeland IJ, Berry JD, Ayers CR, Rohatgi A, Das SR, Khera A, McGuire DK, de Lemos JA, Turer AT. The relationship of body mass and fat distribution with incident hypertension: observations from the Dallas Heart Study. J Am Coll Cardiol. 2014 Sep 9;64(10):997-1002. doi: 10.1016/j.jacc.2014.05.057. PMID 25190234
- [Background] Hutley L, Prins JB. Fat as an endocrine organ: relationship to the metabolic syndrome. Am J Med Sci. 2005 Dec;330(6):280-9. doi: 10.1097/00000441-200512000-00005. PMID 16355012
- [Background] Li P, Liu B, Wu X, Lu Y, Qiu M, Shen Y, Tian Y, Liu C, Chen X, Yang C, Deng M, Wang Y, Gu J, Su Z, Chen X, Zhao K, Sheng Y, Zhang S, Sun W, Kong X. Perirenal adipose afferent nerves sustain pathological high blood pressure in rats. Nat Commun. 2022 Jun 6;13(1):3130. doi: 10.1038/s41467-022-30868-6. PMID 35668093